CLINICAL TRIAL: NCT01709695
Title: Neurobiological Basis of Response to Guanfacine Extended Release in Children and Adolescents With Attention-deficit/Hyperactivity Disorder (ADHD): an Functional Magnetic Resonance Imaging(fMRI) Study of Brain Activation Pre and Post Treatment
Brief Title: Neurobiological Basis of Response to Guanfacine Extended Release in Children and Adolescents With ADHD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Jeffrey Newcorn, Principal Investigator, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 09-1825; HSM:10-00415
Record Dates: First submitted 2012-08-30; First posted 2012-10-18 (Estimated); Results first posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-01

CONDITIONS: ADHD; Attention Deficit Hyperactivity Disorder
Keywords: Intuniv; Attention Deficit Hyperactivity Disorder; fMRI
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- guanfacine hydrochloride XR (Experimental): Flexible dose titration of guanfacine extended release (Intuniv; active medication). The medication is titrated in doses from 1 - 4 mg once daily
  Interventions: Drug: Guanfacine Hydrochloride XR
- Placebo Group (Placebo Comparator): Flexible dose titration of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Guanfacine Hydrochloride XR — Weekly adjustments based on parent ratings of symptoms, side effects, and health status per vital signs up to 4mg maximum dose
  Other Names: INTUNIV non-stimulant medication; GXR
  Arms: guanfacine hydrochloride XR
Drug: Placebo — Weekly adjustments based on parent ratings of symptoms, side effects, and health status per vital signs up to 4mg maximum dose
  Arms: Placebo Group

SUMMARY:
This study proposes to evaluate the effects of guanfacine extended release on brain activation during fMRI in children and adolescents with ADHD between the ages 8-15 and ADHD subjects randomized to placebo treatment.

This study also proposes to collect DNA on study participants, to examine the genetic underpinning of the observed fMRI activation profiles at baseline and in response to treatment. The purpose is to examine polymorphisms of the adrenergic 2A gene (and other related targets) for genetic biomarkers in association with the fMRI findings of this study.

DETAILED DESCRIPTION:
This study proposes to evaluate the effects of guanfacine on brain activation during fMRI in 12 children and adolescents ages 8 - 15 with ADHD treated with once-daily INTUNIV(TM) (guanfacine; GXR) extended release tablets and 12 ADHD subjects randomized to placebo treatment. Children will be comprehensively assessed using a variety of clinical and neuropsychological measures. They will be scanned at baseline while performing both the go/no-go task (a well validated task for measuring inhibitory control (Durston et al., 2002, 2003)) and the Stay Alert task - a new task designed to measure the arousal component of attention, which was used successfully in a recent fMRI study of guanfacine in healthy adults (Clerkin et al., 2009). They will then be treated with GXR or placebo for 6 - 8 weeks in accordance with titration and dosing strategies used in recent Phase III dose optimization trials (e.g., up to 4 mg/day), and re-scanned while performing the same two tasks. The fMRI scans will be conducted using a dedicated research 3.0 T Siemens scanner.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of any subtype of ADHD
* Normal findings on physical exam, laboratory studies, vital signs, and ECG
* Weight = 60 kgs or less
* Able to complete study procedures and swallow capsules;
* Willing to commit to the entire visit schedule
* Off treatment or have been discontinued from their previous medication for two weeks.

Exclusion Criteria:

* Psychiatric comorbidity except Oppositional Defiant Disorder [ODD], Simple Phobia, and dysthymia (unless ongoing medication treatment is required);
* Currently a suicide risk, has previously made a suicide attempt or has a prior history of suicidal behavior;
* Has failed treatment with an adequate trial of an alpha-2 adrenergic agonist;
* Known or suspected allergy, hypersensitivity, or clinically significant intolerance to guanfacine hydrochloride.

Children may not:

* be treated with systemic medication for a medical or psychiatric illness that have CNS effects or affect cognitive function;
* have a known history or presence of structural cardiac abnormalities, exercise-related cardiac events, or clinically significant bradycardia;
* have orthostatic hypotension or a known history of hypertension;
* have an abnormal ECG that is deemed clinically significant;
* have a history of alcohol or other substance abuse or dependence within the last 6 months;
* use any medications that affect BP or heart rate (excluding the subject's current ADHD medication at screening);
* use another investigational medicinal product or participation in a clinical study within 30 days prior to the baseline visit;
* be significantly overweight based on Center for Disease Control and Prevention Body Mass Index (BMI)-for-age gender specific charts;
* have body weight of less than 25kg;
* have a clinically important abnormality on urine drug and alcohol screen (excluding the subject's current ADHD stimulant, if applicable);
* be female and currently pregnant or lactating;
* have symptoms indicative of a primary sleep disorder.
* have braces or other metal permanently placed within their body.
* be too anxious to tolerate the fMRI procedure, or be claustrophobic.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Newcorn, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Result] Bedard AC, Schulz KP, Krone B, Pedraza J, Duhoux S, Halperin JM, Newcorn JH. Neural mechanisms underlying the therapeutic actions of guanfacine treatment in youth with ADHD: a pilot fMRI study. Psychiatry Res. 2015 Mar 30;231(3):353-6. doi: 10.1016/j.pscychresns.2015.01.012. Epub 2015 Jan 19. PMID 25659477

RESULTS

PARTICIPANT FLOW:
Groups:
- Guanfacine Hydrochloride XR: Flexible dose titration of guanfacine extended release - titrated in doses from 1 - 4 mg once daily
Period: Overall Study
Arm/Group | Guanfacine Hydrochloride XR | Placebo Group
Started | 13 | 14
Completed | 12 | 13
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Data unavailable for one participant in each group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Guanfacine Hydrochloride XR | Placebo Group | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.6 (1.7) | 11.5 (2.5) | 11.1 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 9 | 9 | 18
Full Scale IQ [Mean (Standard Deviation); unit: units on a scale] — Full Scale IQ - People who score generally between 70 and 130 are considered to be within the normal range of IQ functioning, where 100 is the theoretical average. Those scoring 130 and above have significantly greater cognitive resources than the average population, and those scoring 70 and below population have significantly fewer cognitive resources.
  units on a scale | 110.0 (21.6) | 101.8 (13.1) | 105.7 (17.75)
Attention-Deficit/Hyperactivity Disorder (ADHD) subtype [Count of Participants; unit: Participants]
  Combined | 8 | 9 | 17
  Inattentive | 4 | 4 | 8
Comorbid Oppositional Defiant Disorder (ODD) [Count of Participants; unit: Participants] | 7 | 4 | 11
Clinical Global Impressions - Severity scale (CGI-S) [Mean (Standard Deviation); unit: units on a scale] — Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's symptoms at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of symptoms at the time of rating 1, normal, not at all ill; 2, minimally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, very servely ill.
  units on a scale | 4.9 (1.0) | 5.4 (0.9) | 5.2 (0.9)
Prior stimulant treatment [Count of Participants; unit: Participants] | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Go/No-go Task Performance Correct Inhibitions
Description: Measures of go/no-go task performance during functional magnetic resonance imaging. Performance on a go-nogo task inside the scanner.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: percentage correct inhibitions
Arm/Group | Guanfacine Hydrochloride XR | Placebo Group
Number analyzed (Participants) | 12 | 13
percentage correct inhibitions
  Baseline Correct inhibitions | 91 (8) | 89 (10)
  8 Weeks Correct inhibitions | 94 (6) | 92 (7)

2. Primary Outcome: Go/No-go Task Reaction Time
Description: as for outcome 1
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Guanfacine Hydrochloride XR | Placebo Group
Number analyzed (Participants) | 12 | 13
ms
  Baseline Reaction time (RT) | 572 (144) | 543 (99)
  Baseline Reaction time standard deviation (RTSD) | 187 (109) | 165 (76)
  8 weeks Reaction time (RT) | 562 (106) | 550 (107)
  8 weeks Reaction time standard deviation (RTSD) | 184 (93) | 166 (73)

3. Secondary Outcome: Clinical Global Impressions (CGI-I)
Description: Clinical response was the Clinical Global Impression-Improvement scale (CGI-I). Lower CGI-I scores indicate greater improvement (1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6= much worse; 7=very much worse.)
Time Frame: up to 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guanfacine Hydrochloride XR | Placebo Group
Number analyzed (Participants) | 12 | 13
units on a scale | 2.0 (0.7) | 2.9 (1.1)

4. Secondary Outcome: Percentage Change in Atomoxetine Stimulant Side Effects Rating Scale (ASSERS)
Description: Side effects rating scale. Assesses side effects known to occur in prior research using stimulant and non stimulant medications for treatment of ADHD. Scores range from 0 (not present) to 9 (severe side effects) and have been reported in aggregate as sum of severity responses on highest dose. This number is the sum of ASSERS, meaning it is the number and severity of side effects experienced. The percentage change in score from baseline.
Time Frame: up to 8 weeks
Measure: Number; unit: percentage of mean effects improvement
Arm/Group | Guanfacine Hydrochloride XR | Placebo Group
Number analyzed (Participants) | 12 | 13
percentage of mean effects improvement | 78 | 65.18

5. Secondary Outcome: Finger Windows
Description: Neuropsychological assessment: Finger Windows - a measure of spatial working memory. The participant shows memory of a demonstrated visual pattern. The examiner models a given sequence of windows and ask the participant to imitate the sequence by placing their finger through the same windows in the correct order. The total number of correct sequences achieved determines the level of performance.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: correct sequences
Arm/Group | Guanfacine Hydrochloride XR | Placebo Group
Number analyzed (Participants) | 12 | 13
correct sequences
  Finger Windows - F | 12.5 (6.52) | 10.75 (4.63)
  Finger Windows -B | 11.35 (5.45) | 8.00 (5.14)

6. Secondary Outcome: Digit Span
Description: Neuropsychological assessment - Digit Span. The Digit Span test is either conducted verbally or using a computer program. A sequence of numbers is shown or read out to the participant. The participant is then told to repeat the numbers that were shown or read to them. This process continues until the participant can no longer remember either the full sequence of numbers or the correct order. This sequence is also continued until the participant makes an error. The Digit Span test is scored by the amount of numbers the participant was able to remember in each test. The scorer must add the total number of correct sequences, backwards and forwards. This test is also scored differently for a range of ages.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: correct sequences
Arm/Group | Guanfacine Hydrochloride XR | Placebo Group
Number analyzed (Participants) | 12 | 13
correct sequences
  Digit Span - F | 6.92 (1.73) | 7.54 (2.54)
  Digit Span - B | 48.62 (8.76) | 48.62 (8.76)

7. Secondary Outcome: Attention Deficit Hyperactivity Disorder Rating Scale IV (ADHDRS IV)
Description: Norm referenced parent interview to assess severity and frequency of ADHD symptoms. Scores are reported as sums 0 (no symptoms) to 54 (severe).
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guanfacine Hydrochloride XR | Placebo Group
Number analyzed (Participants) | 12 | 13
units on a scale
  Baseline | 36.67 (9.01) | 39.15 (9.08)
  End of treatment at 8 weeks | 9.42 (6.96) | 22.69 (11.90)

8. Secondary Outcome: Continuous Performance Test - Commissions
Description: Neuropsychological assessment - Continuous Performance Test - Commissions. CPT is a task-oriented computerized assessment of attention-related problems. Scores are compared with the normative scores for the age, group and gender of the person being tested. A t-score of 50 is equal to the mean, with higher values indicating more problematic behaviors and lower scores indicating less problematic behaviors.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: t-scores
Arm/Group | Guanfacine Hydrochloride XR | Placebo Group
Number analyzed (Participants) | 12 | 13
t-scores | 48.62 (3.81) | 46.99 (2.99)

9. Primary Outcome: Go/No-go Task Performance Correct Responses
Description: as for outcome 1
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: percentage correct responses
Arm/Group | Guanfacine Hydrochloride XR | Placebo Group
Number analyzed (Participants) | 12 | 13
percentage correct responses
  Baseline Correct responses | 76 (18) | 75 (14)
  8 Weeks Correct responses | 79 (15) | 74 (15)

ADVERSE EVENTS:
Arm/Group | Guanfacine Hydrochloride XR | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 4/12 | 3/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Guanfacine Hydrochloride XR (N=12) | Placebo Group (N=13)
Somnolence (General disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Irritability (Psychiatric disorders) | 1 | 1
Increased Anxiety/Panic (Psychiatric disorders) | 0 | 1
Sleepiness (General disorders) | 2 | 2
Irritable and Moody (Psychiatric disorders) | 0 | 2
Difficulty Sleeping (General disorders) | 0 | 1
Viral Infection (Infections and infestations) | 0 | 1 — Sore throat and nasal congestions secondary to common cold
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dizziness upon standing (General disorders) | 1 | 0
Drowsiness (General disorders) | 3 | 0
Appearing sedated (General disorders) | 1 | 0 — could not tolerate dose rise, dose reduced
Aggression (General disorders) | 1 | 0
Tired (General disorders) | 1 | 0
Headache (General disorders) | 1 | 0
Weakness (General disorders) | 1 | 0 — subjective feeling of weakness, without loss of strength.

LIMITATIONS AND CAVEATS:
The small sample size in this pilot study limited power to detect large-sized effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No